CLINICAL TRIAL: NCT03737214
Title: A Multi-center, Open-label, Uncontrolled, Single-arm, Extension Study to Determine the Long-term Safety and Tolerability of Oral Lucerastat in Adult Subjects With Fabry Disease
Brief Title: A Study to Evaluate the Long-term Safety and Tolerability of Lucerastat in Adult Subjects With Fabry Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID-069A302; 2024-513884-20-00 (EU CTIS Number); 2018-002210-12 (EudraCT Number)
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-06

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — migalastat

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label, uncontrolled, single-arm, extension study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lucerastat (Experimental): Dose will be based on subject's eGFR.
  Interventions: Drug: Lucerastat

INTERVENTIONS:
Drug: Lucerastat — Administered in hard gelatin capsules containing 250 mg of lucerastat.

SUMMARY:
A study to determine the long-term safety and tolerability of oral lucerastat in adult subjects with Fabry disease. This study includes a sub-study evaluating kidney Gb3 inclusions (and other histologic lesions) in male participants with classic Fabry disease who have been treated for at least 2 years with lucerastat monotherapy in study ID-069A302.

DETAILED DESCRIPTION:
Study ID-069A302 will continue at each site until lucerastat is commercially available in the respective country, or until all subjects have (prematurely) discontinued the trial, or until the sponsor terminates the study, whichever is earliest.

Note that, in Europe (local protocol amendment), the maximum individual study participation is up to Month 96.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF prior to any study-mandated procedure;
* Subject completed the 6-month, double-blind treatment period in study ID 069A301
* Woman of childbearing potential only if agreement 1) to follow a specified contraception scheme, 2) to undertake monthly urine pregnancy tests.
* Fertile male only if agreement 1) to use a condom, 2) to not father a child.

Exclusion Criteria:

* Pregnant / planning to be become pregnant or lactating subject;
* Subject considered to be at high risk of developing clinical signs of organ involvement within the time period of the study, as per investigator judgment;
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results as per investigator judgment.

In addition, the subject must not be enrolled in study ID-069A302 if at any time during study ID-069A301, one of the following criteria was met:

* Subject's eGFR per the Chronic Kidney Disease Epidemiology Collaboration creatinine equation < 15 mL/min/1.73 m2;
* Subject experienced an event of acute kidney injury Common Terminology Criteria for Adverse Event (CTCAE) grade 2 or above;
* Subject experienced an event of stroke CTCAE grade 3 or above;
* Subject experienced an event of heart failure leading to in-patient hospitalization or prolongation of ongoing hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (AEs) | From enrollment to Follow-up 1 (FU1) visit; duration: for up to 10 years including 1 month Follow-up

OTHER OUTCOMES:
Treatment-emergent serious adverse events (SAEs) | From enrollment to Follow-up 1 (FU1) visit; duration: for up to 10 years including 1 month Follow-up
Subject estimated glomerular filtration rate (eGFR) slope | From baseline to Month 24, Month 48 and Month 72 (duration: up to 6 years)
Change in left ventricular mass index (LVMI) | From baseline to Month 24, Month 48 and Month 72 (duration: up to 6 years)
Change in plasma globotriaosylceramide (Gb3) | From baseline to Month 24, Month 48 and Month 72 (duration: up to 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (42):
- United States (14):
  - University of Alabama at Birmingham - Nephrology Research Clinic, Birmingham, Alabama
  - University of California Irvine, Irvine, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Florida Clinical and Translational Science Institute, UF Clinical Research Center, Gainesville, Florida
  - Rush University Medical Center - Dept of Pediatrics, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital - Division of Medical Genetics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Infusion Associates, Grand Rapids, Michigan
  - University of Pennsylvania - Dept of Medicine, Philadelphia, Pennsylvania
  - Greenwood Genetics Center, Greenville, South Carolina
  - Renal Disease Research Institute LLC, Dallas, Texas
  - Baylore University Medical Center, Dallas, Texas
  - University of Utah - Division of Medical Genetics, Clinical Genetics Research, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia
- Australia (2):
  - Royal Perth Hospital, Department of Nephrology, Perth, Perth
  - Royal Melbourne Hospital - Department of Nephrology, Parkville
- Medizinische Universität Wien, Universitätsklinik für Innere Medizin III, Klinische Abteilung für Nephrologie und Dialyse, Vienna, Austria
- Belgium (2):
  - University Hospital Ghent (UZ Ghent), Ghent
  - University Hospital Gasthuisberg, Leuven (UZ Leuven), Leuven
- Canada (5):
  - University of Calgary - Heritage Medical Research Clinic, Calgary
  - London Health Sciences CTR, Victoria Hospital, London
  - Research Center, Hôpital du Sacré-Coeur de Montréal, Montreal
  - Vancouver General Hospital - Adult Metabolic Diseases Clinic, Vancouver
  - Children's Hospital Research Institute of Manitoba, Winnipeg
- Raymond Poincaré Hosp - Med Genetics Dept, Garches, France
- Germany (4):
  - Universitätsmedizin Berlin - Charité Campus Mitte, Berlin
  - SphinCS GmbH, Höchheim
  - Nephrologicum Markgräflerland MVZ GmbH, Müllheim
  - Universitätsklinikum Würzburg, Würzburg
- Hospital Academisch Medisch Centrum - Department of Internal Medicine, Div. Endrocrinology and Metabolism, Amsterdam, Netherlands
- Haukeland University Hospital, Bergen, Norway
- Poland (3):
  - Clinic of Immunological Diseases and Blood Coagulability Cracow University Hospital, Krakow
  - Narodowy Instytut Kardiologii Stefana kardynała Wyszyńskiego - Państwowy Instytut Badawczy, Warsaw
  - The Children's Memorial Health Institute, Department of Pediatric, Nutrition and Metabolic Diseases, Warsaw
- Spain (4):
  - Vall d'Hebron University Hospital - Unit of Inherited Metabolic Disorders and Rare Diseases, Barcelona
  - Hospital Universitari de Bellvitge / Nephrology Dpt, Barcelona
  - Hospital Universitario Ramon y Cajal. Servicio de Medicina Interna, Madrid
  - Hospital Quironsalud Zaragoza, Zaragoza
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland
- United Kingdom (3):
  - Royal Free London NHS Foundation Trust Lysosomal Storage Disorder Unit; Department of Hematology, London
  - National Hospital for Neurology and Neurosurgery, London
  - Salford Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wanner C, Kimonis V, Politei J, Warnock DG, Uceyler N, Frey A, Cornelisse P, Hughes D. Understanding and modifying Fabry disease: Rationale and design of a pivotal Phase 3 study and results from a patient-reported outcome validation study. Mol Genet Metab Rep. 2022 Mar 26;31:100862. doi: 10.1016/j.ymgmr.2022.100862. eCollection 2022 Jun. PMID 35782623